CLINICAL TRIAL: NCT07194733
Title: Supporting VETerans With Kidney Disease Through Food As Medicine: the Community-based VET FAM Study
Brief Title: Supporting VETerans With Kidney Disease Through Food As Medicine
Acronym: VETFAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: Food Bank of the Rockies (Unknown); National Kidney Foundation, United States (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-1288
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Kidney Diseases; Food/Nutrition Insecurity; Diabetes; Hypertension
MeSH Terms: conditions — Kidney Diseases; Diabetes Mellitus; Hypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VET FAM Product Box and Nutrition Education (Experimental): Veterans with kidney disease stages 3b-4 will receive weekly produce boxes through the Food Bank of the Rockies Food for Health program. Boxes include fresh/canned fruits, vegetables, and other items. Participants will also receive nutrition education materials and brief support to encourage preparation and consumption of the provided foods over the study period.
  Interventions: Other: VET FAM Product Box and Nutrition Education

INTERVENTIONS:
Other: VET FAM Product Box and Nutrition Education — Food boxes and nutrition education

SUMMARY:
The goal of this pilot clinical trial is primarily learn if produce boxes improve clinical outcomes among Veterans with kidney disease and food or nutrition insecurity. Secondly, the study will capture Veterans qualitative perspectives, experience, and engagement through semi-structured interviews.

DETAILED DESCRIPTION:
This study aims to address kidney health disparities by implementing and evaluating a Food is/as Medicine intervention tailored for up to 20 Veterans with CKD. These community-engaged efforts seek to better understand the interrelation of nutrition, health, and socioeconomic factors affecting kidney related or patient-centered, along with quantitative clinical, outcomes. The long-term goal of this work is to develop and demonstrate community-based interventions or efforts that improve dietary adherence/quality, reduce food insecurity, improve nutrition security, and enhance kidney health outcomes while providing sustainability, scalable insights for broader public/kidney health and VA healthcare policies or programs.

Objectives:

Objective 1: Evaluate the short-term impact of culturally and medically tailored food boxes and produce (3-month mid-point):

* Understand Veterans' perceptions of food access, intervention acceptability, education effectiveness, and dietary challenges through semi-structured interviews.
* Investigate participant satisfaction, perceived barriers, and facilitators within the food box program and towards healthy/kidney diet adherence or practices.
* Examine Veterans' nutrition security status and quality of life from baseline to 3-months.

Objective 2: Assess the longitudinal impact and perceived future long-term impact of food boxes (6- month endpoint):

* Investigate Veterans' long-term program experiences, perspectives, satisfaction, and preferences.
* Understand participant confidence, self-efficacy, ability to sustain dietary habits, plans and resources needed post-intervention.
* Examine Veterans' nutrition security status and quality of life from baseline, 3-months, to 6-months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* CKD stage 3b or 4
* Positive screen for nutrition insecurity (e.g., Tufts screener)
* Receiving care at the VA and residing in Food Bank of the Rockies service area
* Ability to provide informed consent, English

Exclusion Criteria:

* Stage 1-3a CKD and stage 5 CKD/ESRD (dialysis or transplant)
* Currently enrolled in a conflicting dietary trial
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Systolic Blood Pressure | Baseline (0-months), 3-months, and 6-months
  Systolic Blood Pressure

SECONDARY OUTCOMES:
Creatinine | Baseline (0-months), 3-months, 6-months
  Measure of kidney function
Estimated Glomerular Filtration Rate (eGFR) | Baseline (0-months), 3-months, and 6-months
  Measure of kidney function
Blood urea nitrogen (BUN) | Baseline (0-months), 3-months, 6-months
  A waster product formed from protein breakdown, also filtered by the kidneys
Albumin | Baseline (0-months), 3-months, 6-months
  A protein that may indication kidney damage, inflammation, nutritional status or other measures
HbA1c | Baseline (0-months), 3-months, and 6-months
  Glycosylated hemoglobin A1c
Kidney disease quality of life (KDQOL) | Baseline (0-months), 3-months, 6-months
  Kidney disease quality of life measured by the KDQOL short form instrument

OTHER OUTCOMES:
Qualitative participant perspectives, experiences, and engagement themes | 3-months and 6-months
  Qualitative semi-structured recorded interviews capturing participant perspectives for themes.

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Perez, PhD, RD, Principal Investigator — US Department of Veterans Affairs
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Veterans Affairs data may only be shared with VA approved investigators and per VA policy.